CLINICAL TRIAL: NCT03084471
Title: An Open-Label, Multi-Centre, Safety Study of Fixed-Dose Durvalumab + Tremelimumab Combination Therapy or Durvalumab Monotherapy in Advanced Solid Malignancies.
Brief Title: An Open-Label, Multi-Centre, Study to Assess the Safety of Fixed-Dose Durvalumab + Tremelimumab Combination Therapy or Durvalumab Monotherapy in Advanced Solid Malignancies.
Acronym: STRONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00068
Record Dates: First submitted 2017-03-07; First posted 2017-03-21 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Malignancies
Keywords: Programmed death ligand 1 (PD-L1); Cytotoxic T-lymphocyte antigen-4 (CTLA-4); Durvalumab in combination with tremelimumab
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12 | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination therapy (Experimental): Combination therapy (durvalumab + tremelimumab) : Patients will receive the combination therapy followed by monotherapy via intravenous (IV) infusion once Q4W:
  * Durvalumab 1,500 mg + tremelimumab 75 mg on Week 0, for up to a maximum of 4 doses (or cycles) and
  * Durvalumab 1,500 mg starting 4 weeks after the last infusion of the combination or discontinuation of tremelimumab.
  Interventions: Biological: MEDI4736 (Durvalumab); Biological: MEDI4736 (Durvalumab) + Tremelimumab
- Monotherapy (Experimental): Monotherapy (Durvalumab 1,500 mg): Patients will receive durvalumab 1,500 mg via IV infusion Q4W on Week 0.
  Interventions: Biological: MEDI4736 (Durvalumab)

INTERVENTIONS:
Biological: MEDI4736 (Durvalumab) — A human monoclonal antibody (mAb) of the immunoglobulin G (IgG) 1 kappa subclass that blocks the interaction of PD-L1 (but not programmed cell death ligand-2) with PD-1 on T cells and CD80 (B7.1) on immune cells (IC).
Biological: MEDI4736 (Durvalumab) + Tremelimumab — Durvalumab: A human mAb of IgG 1 kappa subclass that blocks the interaction of PD-L1 (but not programmed cell death ligand-2) with PD-1 on T cells and CD80 (B7.1) on IC.
  Tremelimumab: A human Ig G2 mAb that completely blocks the interaction of human CTLA-4 (cluster of differentiation [CD]152) with CD80 and CD86 and increase release of cytokines (interleukin [IL]-2 and interferon [IFN]-γ) from human T cells, peripheral blood mononuclear cells and whole blood.
  Arms: Combination therapy

SUMMARY:
To evaluate the safety, tolerability, and anti-tumor activity of the combination of durvalumab + tremelimumab or durvalumab alone in different solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, study to determine the short and long term safety of fixed doses of durvalumab 1500 mg + tremelimumab 75 mg combination therapy or durvalumab 1500 mg monotherapy in patients with advanced solid malignancies. This study is modular in design, one or more of the modules will be opened in a given country / region based on local patient population prevalence, and results of feasibility studies. The total number of patients to be enrolled overall and in each module will depend on the types and number of tumor modules added to the main study and country-specific ancillary studies. The number of patients and sites to be involved in individual countries will be dependent on each module or ancillary study. This study consisted of a screening period, a treatment period, a 90 day safety follow-up period and a survival follow-up period. Patients will receive the investigation product (IP) via intravenous (IV) infusion once every 4 weeks (Q4W) in combination therapy or monotherapy as mentioned below - Combination therapy: Durvalumab 1,500 mg + tremelimumab 75 mg on Week 0, for up to a maximum of 4 doses (or cycles) followed by durvalumab 1,500 mg starting 4 weeks after the last infusion of the combination or discontinuation of tremelimumab.

Monotherapy: Durvalumab 1,500 mg on week 0.

Patients will attend a safety follow-up visit 90 days after study treatment discontinuation. Thereafter, patients will be contacted by phone or electronic communication every 3 months for survival status up to 5 years following date of first patient treatment initiation. All patients will be followed for a minimum of 6 months following enrolment of last patient. It is anticipated that the total enrolment period for the overall study will be approximately 2 to 3 years, with an overall duration of approximately 5 years

ELIGIBILITY:
Inclusion criteria:

1. Must have a life expectancy of at least 12 weeks.
2. Age ≥18 years at the time of screening. For patients aged <20 years and enrolled in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative
3. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations. For patients aged <20 years and enrolling in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative.
4. Disease not amenable to curative surgery
5. Eastern Cooperative Oncology Group (ECOG) performance status as defined in the specific module.
6. Body weight >30 kg.
7. No prior exposure to anti-PD-1 or anti-PD-L1, including on another AstraZeneca study. Exposure to other investigational agents may be permitted after discussion with the Sponsor.
8. Adequate organ and marrow function as defined below

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count ≥1.0 × 109 /L
   * Platelet count ≥75 × 109/L
   * Serum bilirubin ≤1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.
   * ALT and AST ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN
   * Measured creatinine clearance (CL) >40 mL/min or calculated creatinine clearance (CL) >40 mL/min as determined by Cockcroft-Gault (using actual body weight)

   Males:

   Creatinine CL = Weight (kg) × (140 - Age) (mL/min) 72 × serum creatinine (mg/dL)

   Females:

   Creatinine CL = Weight (kg) × (140 - Age) x 0.85 (mL/min) 72 × serum creatinine (mg/dL)
9. Female patients of childbearing potential (ie, not surgically sterile or post menopausal) who are sexually active with a non sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy (see Section 3.8 and specifically Table 1).
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test (per Section 4) for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
11. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle- stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Non sterilized male patients who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 180 days after receipt of the final dose of durvalumab + tremelimumab combination therapy or 90 days after receipt of the final dose of durvalumab monotherapy.

Exclusion criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous IP assignment in the present study.
3. Concurrent enrollment in another clinical study, or another sub-study of this protocol, unless it is an observational (non-interventional) clinical study or during the follow up period of an interventional study.
4. Participation in another clinical study with an investigational product during the last 28 days or 5 half-lives, whichever is longer, prior to the first dose of study treatment.
5. Any concurrent chemotherapy, investigational agent, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
6. Local treatment of isolated lesions for palliative intent is acceptable (eg, local surgery or radiotherapy).
7. Receipt of any investigational anticancer therapy within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study treatment.
8. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable.
9. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
10. History of allogenic organ transplantation.
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, ILD, serious chronic GI conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of investigational product (durvalumab + tremelimumab) and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis
14. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on baseline brain imaging (please refer to RECIST for details on the imaging modality) obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least 4 weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10 mg/day of prednisone or its equivalent and anti-convulsants for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
15. History of active primary immunodeficiency.
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
18. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
19. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
20. Known allergy or hypersensitivity to study drug(s) or compounds of similar biologic composition to the study drug(s), or any of the study drug excipients.
21. Any unresolved NCI CTCAE Grade ≥2 toxicities from prior anti cancer therapy with the exception of vitiligo, alopecia, and the laboratory values defined in the inclusion criteria.

    * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician
22. For women only, currently pregnant (confirmed with positive pregnancy test) or breast feeding.
23. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy.
24. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (10):
  - Research Site, Santa Rosa, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tinley Park, Illinois
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, East Setauket, New York
  - Research Site, Greenville, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Blacksburg, Virginia
  - Research Site, Spokane, Washington
- Canada (9):
  - Research Site, Moncton, New Brunswick
  - Research Site, Brampton, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Québec, Quebec
- France (19):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Gütersloh
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, Münster
  - Research Site, Stuttgart
  - Research Site, Würzburg
- Italy (15):
  - Research Site, Ancona
  - Research Site, Arezzo
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Lecce
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Udine
- Research Site, Leiden, Netherlands
- South Korea (3):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Seoul
- United Kingdom (3):
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Sonpavde GP, Sternberg CN, Loriot Y, Marabelle A, Lee JL, Flechon A, Roubaud G, Pouessel D, Zagonel V, Calabro F, Banna GL, Shin SJ, Vera-Badillo FE, Powles T, Hellmis E, Miranda PAP, Lima AR, Emeribe U, Oh SM, Hotte SJ. Primary results of STRONG: An open-label, multicenter, phase 3b study of fixed-dose durvalumab monotherapy in previously treated patients with urinary tract carcinoma. Eur J Cancer. 2022 Mar;163:55-65. doi: 10.1016/j.ejca.2021.12.012. Epub 2022 Jan 15. PMID 35042068
- See also: redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191C00068&attachmentIdentifier=67484637-c120-4784-9f00-aae6e369b5f2&fileName=D4191C00068_CSP_redacted.pdf&versionIdentifier=
- See also: redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191C00068&attachmentIdentifier=8e9421af-9880-4525-a031-c1e541b74a5c&fileName=D4191C00068_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and none of the exclusion criteria were randomized at 77 study centers across 8 countries (Canada, France, Germany, Italy, Republic of Korea, Netherlands, United Kingdom and United States of America).
Pre-assignment Details: During the screening period (4 weeks), eligible participants signed the informed consent. All the study assessments were performed as per the schedule of assessment.
Groups:
- Durvalumab: All participants received fixed-dose of durvalumab 1500 mg every 4 weeks until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Durvalumab
Started | 867
Completed | 0
Not Completed | 867
Not completed — Development of study specific discontinuation criteria | 2
Not completed — Condition under investigation worsened | 84
Not completed — Lack of therapeutic response | 2
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 73
Not completed — Withdrawal by Subject | 12
Not completed — Disease relapse | 181
Not completed — Subjective disease progression | 359
Not completed — Other (as recorded) | 33
Not completed — Patients who were still on study treatment at Data Cutoff | 120

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab
Number analyzed (Participants) | 867
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 694
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was not a mandatory variable to be collected in some sites due to data privacy reasons. Hence, the total number of participants analysed for race is lesser than Overall (Safety Analysis Set)
  Participants
    number analyzed (Participants) | 603
    American Indian or Alaska Native | 0
    Asian | 65
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 508
    More than one race | 0
    Unknown or Not Reported | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Incidence, severity, nature, seriousness, intervention/treatment, outcome, and causality of AESIs were assessed. AESIs included events with a potential inflammatory or immune-mediated mechanism that required interventions such as steroids, immunosuppressants, and/or hormone replacement therapy.
Time Frame: From screening to safety follow up visit (90 days after last dose), up to approximately 3 years.
Population: Safety analysis set: all enrolled participants who received at least one dose of durvalumab.
Measure: Number; unit: participants
Groups:
- AESI: AESIs are defined as AEs with a likely inflammatory or immune-mediated pathophysiological basis, resulting from the mechanism of action of durvalumab and/or tremelimumab and requiring more frequent monitoring and/or interventions, such as corticosteroids, immunosuppressants, and/or endocrine therapy.
- AEPI: AEPIs are defined as AEs that could have a potential inflammatory or immune-mediated pathophysiological basis, resulting from the mechanism of action of durvalumab but are more likely to have occurred due to other pathophysiological mechanisms, thus, the likelihood of the event being inflammatory or immune-mediated in nature is not high and/or is most often or usually explained by the other causes.
- imAE: The imAEs that occurred during this study were determined by a programmatic algorithm that required specific treatment for AESIs to be considered imAEs; the same specific treatment was required for AEPIs as well.
Arm/Group | AESI | AEPI | imAE
Number analyzed (Participants) | 867 | 867 | 867
participants
  Any adverse event (AE) | 265 | 300 | 97
  Any AE of common terminology criteria for AEs Grade 3 or 4 | 21 | 49 | 17
  Any serious adverse event (SAE) (including events with outcome = death) | 19 | 13 | 11
  Any AE with outcome = death | 1 | 0 | 0
  Any AE, causally related to treatment | 191 | 145 | 87
  Any AE of common terminology criteria Grade 3 or 4, causally related to treatment | 15 | 20 | 16
  Any SAE, causally related to treatment | 14 | 3 | 10
  Any AE with outcome = death, causally related to treatment | 1 | 0 | 0
  Any AE leading to discontinuation of study treatment | 12 | 7 | 10
  Event outcome resolved | 140 | 119 | 32
  Event outcome not resolved | 124 | 181 | 65

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first date of treatment until death due to any cause.
Time Frame: From screening to final data cutoff (maximum up to 4 years) following date of first patient treatment initiation.
Population: Safety analysis set: all enrolled participants who received at least 1 dose of durvalumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab
Number analyzed (Participants) | 867
months | 7.0 [6.44 to 8.18]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Incidence, severity, nature, seriousness, intervention/treatment, outcome, and causality of treatment-emergent AEs (including SAEs) will be assessed
Time Frame: From screening to safety follow up visit (90 days after last dose), maximum up to 4 years.
Population: Safety analysis set: all enrolled participants who received at least one dose of durvalumab.
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 867
participants
  Any AE | 787
  Any AE causally related to any study treatment | 407
  Any AE of common terminology criteria grade 3 or higher | 365
  Any AE of common terminology criteria grade 3 or higher, causally related to study treatment | 78
  Any AE with outcome = death | 42
  Any AE with outcome = death causally related to study treatment | 9
  Any SAE (including events with outcome = death) | 254
  Any SAE (including events with outcome = death) causally related to study treatment | 41
  Any AE leading to discontinuation of study treatment | 77
  Any AE leading to discontinuation of study treatment causally related to study treatment | 33

ADVERSE EVENTS:
Time Frame: From screening to safety follow up visit (90 days after last dose), maximum up to 4 years.
Description: MedDRA version 23.0
Arm/Group | Durvalumab
All-Cause Mortality (participants affected / at risk) | 600/867
Serious Adverse Events (participants affected / at risk) | 254/867
Other Adverse Events (participants affected / at risk) | 669/867
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab (N=867)
Sepsis (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 17
Pyelonephritis (Infections and infestations) | 8
Device related infection (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 6
Urosepsis (Infections and infestations) | 5
Pyelonephritis acute (Infections and infestations) | 4
Bacterial infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Atypical pneumonia (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Clostridium colitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Enterobacter sepsis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Fournier's gangrene (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1
Spinal cord infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal atony (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 8
Haematuria (Renal and urinary disorders) | 7
Renal failure (Renal and urinary disorders) | 4
Hydronephrosis (Renal and urinary disorders) | 3
Urinary tract obstruction (Renal and urinary disorders) | 3
Urinary tract inflammation (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urine abnormality (Renal and urinary disorders) | 1
Tumour hyperprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
General physical health deterioration (General disorders) | 7
Death (General disorders) | 5
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Drug intolerance (General disorders) | 1
Generalised oedema (General disorders) | 1
Hyperthermia (General disorders) | 1
Hyperthermia malignant (General disorders) | 1
Performance status decreased (General disorders) | 1
Vascular stent thrombosis (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Stomal hernia (Injury, poisoning and procedural complications) | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Basilar artery occlusion (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Frontal lobe epilepsy (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
VIth nerve disorder (Nervous system disorders) | 1
Blood creatinine increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Troponin increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Hepatitis (Hepatobiliary disorders) | 2
Hepatocellular injury (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Device occlusion (Product Issues) | 2
Device dislocation (Product Issues) | 1
Stent malfunction (Product Issues) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Scrotal mass (Reproductive system and breast disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab (N=867)
Asthenia (General disorders) | 228
Fatigue (General disorders) | 83
Pyrexia (General disorders) | 79
Oedema peripheral (General disorders) | 75
Constipation (Gastrointestinal disorders) | 171
Diarrhoea (Gastrointestinal disorders) | 136
Nausea (Gastrointestinal disorders) | 126
Vomiting (Gastrointestinal disorders) | 76
Abdominal pain (Gastrointestinal disorders) | 64
Anaemia (Blood and lymphatic system disorders) | 172
Decreased appetite (Metabolism and nutrition disorders) | 149
Cough (Respiratory, thoracic and mediastinal disorders) | 84
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 74
Back pain (Musculoskeletal and connective tissue disorders) | 82
Arthralgia (Musculoskeletal and connective tissue disorders) | 65
Pruritus (Skin and subcutaneous tissue disorders) | 109
Blood creatinine increased (Investigations) | 48
Weight decreased (Investigations) | 46
Urinary tract infection (Infections and infestations) | 84
Haematuria (Renal and urinary disorders) | 64
Hypothyroidism (Endocrine disorders) | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure of study information is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03084471/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03084471/SAP_003.pdf